CLINICAL TRIAL: NCT03277729
Title: A Phase I/II Study to Evaluate the Safety of Cellular Immunotherapy Using Autologous T Cells Engineered to Express a CD20-Specific Chimeric Antigen Receptor for Patients With Relapsed or Refractory B Cell Non-Hodgkin Lymphomas
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Mustang Bio (Industry)
Responsible Party: Principal Investigator, Mazyar Shadman, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9738; NCI-2017-01595 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9738 (Other: Fred Hutch/University of Washington Cancer Consortium); RG9217017 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-09

CONDITIONS: Recurrent B-Cell Non-Hodgkin Lymphoma; Recurrent Chronic Lymphocytic Leukemia; Recurrent Diffuse Large B-Cell Lymphoma; Recurrent Follicular Lymphoma; Recurrent Lymphoplasmacytic Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Refractory Diffuse Large B-Cell Lymphoma; Refractory Follicular Lymphoma; Refractory Lymphoplasmacytic Lymphoma; Refractory Mantle Cell Lymphoma; Refractory Transformed Non-Hodgkin Lymphoma; Recurrent Transformed B-Cell Non-Hodgkin Lymphoma; Recurrent Transformed Chronic Lymphocytic Leukemia; Refractory Marginal Zone Lymphoma; Refractory Transformed B-Cell Non-Hodgkin Lymphoma; Refractory Transformed Chronic Lymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Small Lymphocytic Lymphoma; Recurrent Central Nervous System Lymphoma; Refractory Central Nervous System Lymphoma
Keywords: Lymphoid Leukemia; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Leukemia, Lymphoid; Lymphoma, Non-Hodgkin | interventions — Immunotherapy, Adoptive; Cyclophosphamide; Leukapheresis; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CD20-specific CAR T cell, chemotherapy) (Experimental): Patients undergo leukapheresis and may receive treatment after if needed for disease control. Patients then receive cyclophosphamide IV. Patients may also receive fludarabine IV. After 36-96 hours, patients receive CD20-specific CAR T cell infusion IV over 20-30 minutes.
  Interventions: Biological: Chimeric Antigen Receptor T-Cell Therapy; Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Procedure: Leukapheresis; Drug: Fludarabine Phosphate

INTERVENTIONS:
Biological: Chimeric Antigen Receptor T-Cell Therapy — Given CD20 CAR T cell IV
  Other Names: CAR T-cell therapy; CAR T Infusion; CAR T Therapy
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Leukapheresis — Undergo leukapheresis
  Other Names: Leukocytopheresis; Therapeutic Leukopheresis
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara; Fludarabine-5''-Monophosphate; SH T 586

SUMMARY:
The purpose of this research is to find the best dose of genetically modified T-cells, to study the safety of this treatment, and to see how well it works in treating patients with B cell non-Hodgkin lymphoma that has come back (relapsed) or did not respond to previous treatment (refractory).

DETAILED DESCRIPTION:
OUTLINE:

This is a phase I/II dose-escalation study of CD20-specific CAR T cell therapy.

Patients undergo leukapheresis and may receive treatment after if needed for disease control. Patients then receive cyclophosphamide intravenously (IV). Patients may also receive fludarabine IV. After 36-96 hours, patients receive CD20-specific CAR T cell infusion IV over 20-30 minutes.

Patients will be actively participating in the study for approximately 15 months. The total time includes the time for the T cells to be made, the T cell infusion, and for approximately 12 months after the T cell infusion is given. After completion of study treatment, patients are followed up for a minimum of 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have B-cell non-Hodgkin lymphoma or chronic lymphocytic leukemia/small lymphocytic lymphoma. Eligible lymphoma subtypes include (but not limited to): mantle cell, follicular, lymphoplasmacytic, marginal zone, transformed indolent B cell lymphoma (including transformed chronic lymphoid leukemia [CLL]), or diffuse large B cell lymphoma that has relapsed after a response to at least one prior therapy regimen or is refractory to prior therapy; patients with mantle cell lymphoma must have previously been treated with a Bruton tyrosine kinase (BTK) inhibitor and have either had disease progression, intolerance, or exposure to the drug for at least 3 months; patients with CLL/SLL are eligible if they had disease progression or intolerance to BTKis and/or a BCL-2 inhibitors; they are also required to have been treated with the other agent for at least 3 months (i.e. patients with progression/intolerance to BTKi need to be treated with a BCL-2 inhibitor for at least 3 months, and patients with progression/intolerance to BCL-2 inhibitor need at least 3 months of exposure to a BTKi); patients with de novo diffuse large B-cell lymphoma (DLBCL) must meet one of the following criteria:

  * Biopsy-proven refractory disease after a frontline regimen containing both an anthracycline and rituximab or other anti-CD20 antibody (i.e. "primary refractory"), where any disease recurring within 6 months of completion of the regimen is considered refractory
  * Relapsed or refractory disease after at least one of the following:

    * At least 2 lines of therapy (including at least one with an anthracycline and anti-CD20 antibody)
    * Autologous stem cell transplant
    * Allogeneic stem cell transplant
* Patients with large cell lymphoma transformed from indolent lymphomas are eligible if previously treated with anthracycline containing regimen for either the indolent or large cell histology
* Patients with central nervous system (CNS) lymphoma need to meet one of the following criteria:

  * Primary CNS lymphoma:

    * Progressive disease after 3 cycles or an inadequate response after at least 4 cycles of a high-dose methotrexate (MTX) containing regimen in the opinion of the treating physician, OR
    * Not eligible for MTX therapy due to commodities or tolerance issues per treating physician OR
    * Recurrent disease after an initial response to MTX-based treatment
  * Secondary CNS lymphoma:

    * An inadequate rtesponse to at least 2 cycles of a MTX containing regimen, OR
    * Recurrent disease after an initial response to MTX-based treatment
* Patients must be 18 years of age or older, of any gender, race or ethnicity
* Patients must be capable of understanding and providing a written informed consent
* Negative serum pregnancy test within 2 weeks before enrollment for women of childbearing potential, defined as those who have not been surgically sterilized or who have not been free of menses for at least 1 year
* Fertile male and female patients must be willing to use an effective contraceptive method before, during, and for at least 4 months after the CAR T cell infusion
* Patients must have a Karnofsky performance status of >= 60%
* Confirmation of diagnosis by internal pathology review of initial or subsequent biopsy or other pathologic material at Fred Hutchinson Cancer Research Center (FHCRC)/Seattle Cancer Care Alliance (SCCA)/University of Washington (UW)/Harborview Medical Center (HMC)
* Evidence of CD20 expression by immunohistochemistry or flow cytometry on the tumor specimen obtained with the biopsy performed with screening; if the CD20 expression on the screening tumor biopsy is unclear or could not be assessed due to technical reasons, CD20 expression on a concomitant tumor specimen (such as marrow biopsy or circulating tumor cells) may be used to satisfy this requirement. For CLL and lymphoplasmacytic lymphoma/Waldenström macroglobulinemia (WM) patients, the screening tumor biopsy can we waived for clinical reasons after discussion with the study principal investigator (PI). For patients with CNS lymphoma, a screening tumor biopsy is not required and evidence of CD20 expression can be documented from the original or prior biopsies
* Serum creatinine =< 2.5
* Total bilirubin =< 3.0 mg/dL
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 5 x the upper limit of normal
* Adequate pulmonary function, defined as =< grade 1 dyspnea and saturated oxygen (SaO2) >= 92% on room air; if pulmonary function test (PFT)s are performed based on the clinical judgment of the treating physician, patients with forced expiratory volume in 1 second (FEV1) >= 50% of predicted and carbon monoxide diffusing capability (DLCO) (corrected) of >= 40% of predicted will be eligible
* Adequate cardiac function, defined as left ventricular ejection fraction (LVEF) of >= 50% as assessed by echocardiogram or multigated acquisition (MUGA) scan, or LVEF of 45-49% and clearance by a cardiologist
* Measurable disease that can be accurately measured in at least one dimension as >= 1.5 cm with computed tomography (CT), ultrasound, or magnetic resonance imaging (MRI) techniques. Extranodal disease that is measurable by fludeoxyglucose F-18 (FDG)-positron emission tomography (PET) imaging only will also be allowed. Note that if an excisional biopsy was performed that removed the sole site of measurable disease, the patient will not be eligible for leukapheresis and generation of CAR T cell product
* For patients with CNS lymphoma, a lesion >= 1cm on brain or spine MRI is required
* Patients with waldenstrom macroglobulinemia (WM) without radiologic evidence of disease are eligible if they have measurable disease, as defined by serum monoclonal M-spike of >= 0.5 g/dL
* ELIGIBILITY FOR LYMPHODEPLETION CHEMOTHERAPY: Absence of uncontrolled active infection (bacterial, fungal, viral, mycobacterial) not responding to treatment with antibiotics, antiviral agents, or antifungal agents
* ELIGIBILITY FOR LYMPHODEPLETION CHEMOTHERAPY: Absence of active autoimmune disease requiring ongoing systemic immunosuppressive therapy
* ELIGIBILITY FOR LYMPHODEPLETION CHEMOTHERAPY: Negative serum pregnancy test within 2 weeks before lymphodepletion chemotherapy for women of childbearing potential, defined as those who have not been surgically sterilized or who have not been free of menses for at least 1 year
* ELIGIBILITY FOR LYMPHODEPLETION CHEMOTHERAPY: No treatment with any investigational agent on a different clinical trial between enrollment and lymphodepleting chemotherapy
* ELIGIBILITY FOR LYMPHODEPLETION CHEMOTHERAPY: Serum creatinine =< 2.5
* ELIGIBILITY FOR LYMPHODEPLETION CHEMOTHERAPY: Total bilirubin =< 3.0 mg/dL
* ELIGIBILITY FOR LYMPHODEPLETION CHEMOTHERAPY: AST and ALT =< 5 x the upper limit of normal
* ELIGIBILITY FOR LYMPHODEPLETION CHEMOTHERAPY: Adequate pulmonary function, defined as =< grade 1 dyspnea and SaO2 >= 92% on room air; if PFTs are performed based on the clinical judgment of the treating physician, patients with FEV1 >= 50% of predicted and DLCO (corrected) of >= 40% of predicted will be eligible
* ELIGIBILITY FOR LYMPHODEPLETION CHEMOTHERAPY: Adequate cardiac function, defined as left ventricular ejection fraction (LVEF) of >= 50% as assessed by echocardiogram or MUGA scan, or LVEF of 45-49% and clearance by a cardiologist; if subject receives cardiotoxic chemotherapy after enrollment, repeat echocardiogram or MUGA is required to reestablish eligible LVEF
* ELIGIBILITY FOR LYMPHODEPLETION CHEMOTHERAPY: Patients must have a Karnofsky performance status of >= 60%. Patients with CNS lymphoma with KPS of >= 50% are eligible if performance status is low because of the active lymphoma
* ELIGIBILITY FOR LYMPHODEPLETION CHEMOTHERAPY: Measurable disease that can be accurately measured in at least one dimension as >= 1.5 cm with CT, ultrasound, or MRI techniques; extranodal disease that is measurable by FDG-PET imaging only will also be allowed; note that if an excisional biopsy was performed that removed the sole site of measurable disease, the patient is not be eligible for lymphodepletion and CAR T cell infusion; measurable disease can be based on the imaging study done during the screening unless the patient received treatment in the interim, in which case imaging should be repeated. For patients with CNS lymphoma, a lesion >= 1 cm on the brain or spine MRI is required. Patients with WM without radiologic evidence of disease are eligible if they have measurable disease, as defined by serum IgM level >= 0.5g/dL
* ELIGIBILITY FOR LYMPHODEPLETION CHEMOTHERAPY: Patients must require no corticosteroid therapy or dose of less than 15 mg per day of prednisone or the equivalent; pulsed corticosteroid dose for disease control is acceptable until the day before the start of lymphodepletion
* ELIGIBILITY FOR LYMPHODEPLETION CHEMOTHERAPY: Patients must have no active acute or chronic GVHD

Exclusion Criteria:

* Active autoimmune disease requiring systemic immunosuppressive therapy
* Patients requiring corticosteroid therapy at a dose of 15 mg or more per day of prednisone or the equivalent; pulsed corticosteroid dose for disease control is acceptable
* Patients who are human immunodeficiency virus (HIV) seropositive
* Women who are pregnant or breastfeeding
* Significant cardiovascular diseases within the past 6 months including uncontrolled congestive heart failure (> New York Heart Association [NYHA] class II), myocardial infarction, unstable angina, or uncontrolled arrhythmia
* History of severe immediate hypersensitivity reaction to cyclophosphamide or fludarabine
* History or presence of clinically relevant non-lymphoma central nervous system pathology, including seizures that are uncontrolled on anticonvulsant therapy (>= 1 seizure in the last year), paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson disease, cerebellar disease, or psychosis
* Treatment with any investigational agent on a different clinical trial within 4 weeks prior to enrollment, unless the patient is documented to be unresponsive to the therapy and at least 3 half-lives have elapsed prior to enrollment
* Treatment with any anti-CD19 or anti-CD20 antibody or antibody-drug conjugate therapy within 4 weeks before enrollment
* Previous treatment with CD19-targeted CAR T cells that has resulted in ongoing B cell aplasia at the time of enrollment; patients that demonstrate recovery of normal B cells (>= 20 B cells/ul) by flow cytometry at any point 28 days or later after CD19 CAR T cell infusion will be considered to have functional loss of CD19 CAR T cells and are potentially eligible
* Patients with systemic disease without radiologic evidence of CNS involvement and with isolated CSF involvement detectable by flow cytometry are eligible for enrollment in systemic disease cohorts if neurologically asymptomatic. CSF involvement is not an exclusion for patients enrolled as a primary or secondary CNS lymphoma.
* Presence of active acute or chronic graft versus host disease (GVHD)
* Uncontrolled active infection (bacterial, fungal, viral, mycobacterial) not responding to treatment with intravenous antibiotics, antiviral or antifungal agents
* Patients with concurrent known additional malignancy that is progressing and/or requires active treatment; exceptions include squamous or basal cell carcinoma of the skin and low grade prostate carcinoma (Gleason grade =< 6). Maintenance anti-hormone therapies for breast or prostate cancers are allowed and are not considered active treatment
* Patients with blood or platelet transfusion within 1 week prior to signing Consent A, or with platelets < 50,000/mm^3, neutrophils < 750/mm^3, or hemoglobin < 8.5 g/dL, unless the cytopenias are considered by the treating physician to be largely due to marrow involvement by lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2039-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mazyar Shadman, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fifty-three participants were enrolled but three participants did not move on to treatment due to worsening of their disease status. They were not assigned to a treatment dose level.
Groups:
- Dose Level 0 of CD20 CAR T Cells: Patients undergo leukapheresis and may receive treatment after if needed for disease control. Patients then receive cyclophosphamide IV. Patients may also receive fludarabine IV. After 36-96 hours, patients receive CD20-specific CAR T cell infusion IV over 20-30 minutes.
  Arm 1 contains patients treated at Dose Level 0 (1 x 10^5 tCD19+ T cells/kg, CAR T Cell Dose Inclusion Range: 8.51 x 10^4 - 2.80 x 10^5 tCD19+ T cells/kg)
  Chimeric Antigen Receptor T Cell Therapy: CD20 CAR T cell IV
  Leukapheresis: Undergo leukapheresis
  Cyclophosphamide: Given IV
  Fludarabine Phosphate: Given IV
- Dose Level 1 of CD20 CAR T Cells: Patients undergo leukapheresis and may receive treatment after if needed for disease control. Patients then receive cyclophosphamide IV. Patients may also receive fludarabine IV. After 36-96 hours, patients receive CD20-specific CAR T cell infusion IV over 20-30 minutes.
  Arm 2 contains patients treated at Dose Level 1 (3.3 x 10^5 tCD19+ T cells/kg, CAR T Cell Dose Inclusion Range: 2.81 x 10^5 - 8.50 x 10^5 tCD19+ T cells/kg)
  Chimeric Antigen Receptor T Cell Therapy: CD20 CAR T cell IV
  Leukapheresis: Undergo leukapheresis
  Cyclophosphamide: Given IV
  Fludarabine Phosphate: Given IV
- Dose Level 2 of CD20 CAR T Cells: Patients undergo leukapheresis and may receive treatment after if needed for disease control. Patients then receive cyclophosphamide IV. Patients may also receive fludarabine IV. After 36-96 hours, patients receive CD20-specific CAR T cell infusion IV over 20-30 minutes.
  Arm 3 contains patients treated at Dose Level 2 (1 x 10^6 tCD19+ T cells/kg, CAR T Cell Dose Inclusion Range: 8.51 x 10^5 - 2.80 x 10^6 tCD19+ T cells/kg)
  Chimeric Antigen Receptor T Cell Therapy: CD20 CAR T cell IV
  Leukapheresis: Undergo leukapheresis
  Cyclophosphamide: Given IV
  Fludarabine Phosphate: Given IV
- Dose Level 3 of CD20 CAR-T Cells: Patients undergo leukapheresis and may receive treatment after if needed for disease control. Patients then receive cyclophosphamide IV. Patients may also receive fludarabine IV. After 36-96 hours, patients receive CD20-specific CAR T cell infusion IV over 20-30 minutes.
  Arm 4 contains patients treated at Dose Level 3 (3.3 x 10^6 tCD19+ T cells/kg, CAR T Cell Dose Inclusion Range: 2.81 x 10^6 - 8.50 x 10^6 tCD19+ T cells/kg)
  Chimeric Antigen Receptor T Cell Therapy: CD20 CAR T cell IV
  Leukapheresis: Undergo leukapheresis
  Cyclophosphamide: Given IV
  Fludarabine Phosphate: Given IV
- Dose Level 4 of CD20 CAR-T Cells: Patients undergo leukapheresis and may receive treatment after if needed for disease control. Patients then receive cyclophosphamide IV. Patients may also receive fludarabine IV. After 36-96 hours, patients receive CD20-specific CAR T cell infusion IV over 20-30 minutes.
  Arm 5 contains patients treated at Dose Level 4 (1 x 10^7 tCD19+ T cells/kg, CAR T Cell Dose Inclusion Range: > 8.5 x 10^6 tCD19+ T cells/kg)
  Chimeric Antigen Receptor T Cell Therapy: CD20 CAR T cell IV
  Leukapheresis: Undergo leukapheresis
  Cyclophosphamide: Given IV
  Fludarabine Phosphate: Given IV
Period: Overall Study
Arm/Group | Dose Level 0 of CD20 CAR T Cells | Dose Level 1 of CD20 CAR T Cells | Dose Level 2 of CD20 CAR T Cells | Dose Level 3 of CD20 CAR-T Cells | Dose Level 4 of CD20 CAR-T Cells
Started | 1 | 8 | 4 | 6 | 31
Completed | 1 | 1 | 0 | 5 | 20
Not Completed | 0 | 7 | 4 | 1 | 11

BASELINE CHARACTERISTICS:
Population: Patients enrolled and treated on study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 0 of CD20 CAR T Cells | Dose Level 1 of CD20 CAR T Cells | Dose Level 2 of CD20 CAR T Cells | Dose Level 3 of CD20 CAR-T Cells | Dose Level 4 of CD20 CAR-T Cells | Total
Number analyzed (Participants) | 1 | 8 | 4 | 6 | 31 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (0) | 61 (9) | 61 (8) | 59 (9) | 67 (8) | 64 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 1 | 2 | 13 | 19
  Male | 0 | 6 | 3 | 4 | 18 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 1 | 7 | 4 | 6 | 28 | 46
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 8 | 4 | 6 | 31 | 50

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicities (DLT) Rate
Description: Will be graded by Common Terminology Criteria for Adverse Events version 4.0. Observed DLT rates will be summarized based on the DLT-Evaluable analysis set. Outcome reported as count of participants in each arm who experienced a DLT.
Time Frame: Up to 28 days
Measure: Number; unit: participants
Arm/Group | Dose Level 0 of CD20 CAR T Cells | Dose Level 1 of CD20 CAR T Cells | Dose Level 2 of CD20 CAR T Cells | Dose Level 3 of CD20 CAR-T Cells | Dose Level 4 of CD20 CAR-T Cells
Number analyzed (Participants) | 1 | 8 | 4 | 6 | 31
participants | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Complete Remission
Description: Will be assessed based on the Lugano criteria.
Time Frame: Up to 15 years
Reporting Status: Not Posted

3. Secondary Outcome: Progression-free Survival (PFS)
Description: A Cox proportional hazards model will be used to evaluate PFS.
Time Frame: Duration from study enrollment to progression or death due to any cause (whichever comes first), assessed up to 15 years
Reporting Status: Not Posted

4. Secondary Outcome: Overall Survival (OS)
Description: A Cox proportional hazards model will be used to evaluate OS.
Time Frame: Duration from study enrollment to death due to any cause, assessed up to 15 years
Reporting Status: Not Posted

5. Secondary Outcome: Incidence of Adverse Events
Description: Will be assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: Up to 15 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events and All-Cause Mortality were assessed up to 1 year after CAR T-cell infusion. No patients received more than one CAR T cell infusion, so AE assessment period was only 1 year after first and only CAR T infusion for all patients.
Arm/Group | Dose Level 0 of CD20 CAR T Cells | Dose Level 1 of CD20 CAR T Cells | Dose Level 2 of CD20 CAR T Cells | Dose Level 3 of CD20 CAR-T Cells | Dose Level 4 of CD20 CAR-T Cells
All-Cause Mortality (participants affected / at risk) | 0/1 | 2/8 | 3/4 | 3/6 | 7/31
Serious Adverse Events (participants affected / at risk) | 1/1 | 2/8 | 1/4 | 2/6 | 18/31
Other Adverse Events (participants affected / at risk) | 1/1 | 8/8 | 4/4 | 6/6 | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 0 of CD20 CAR T Cells (N=1) | Dose Level 1 of CD20 CAR T Cells (N=8) | Dose Level 2 of CD20 CAR T Cells (N=4) | Dose Level 3 of CD20 CAR-T Cells (N=6) | Dose Level 4 of CD20 CAR-T Cells (N=31)
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 0 | 2 | 12
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 3
Fever (General disorders) | 0 | 0 | 0 | 0 | 5
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Immune system disorders (Immune system disorders) | 0 | 0 | 0 | 0 | 2 — Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
General disorders and administration site conditions - Other, COVID (General disorders) | 0 | 0 | 0 | 0 | 1 — COVID19
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Spasticity (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 0 of CD20 CAR T Cells (N=1) | Dose Level 1 of CD20 CAR T Cells (N=8) | Dose Level 2 of CD20 CAR T Cells (N=4) | Dose Level 3 of CD20 CAR-T Cells (N=6) | Dose Level 4 of CD20 CAR-T Cells (N=31)
Lymphocyte count decreased (Investigations) | 1 | 8 | 4 | 6 | 28
Neutrophil count decreased (Investigations) | 1 | 7 | 4 | 5 | 29
White blood cell decreased (Investigations) | 1 | 8 | 4 | 5 | 28
Anemia (Blood and lymphatic system disorders) | 1 | 6 | 2 | 3 | 25
Fatigue (General disorders) | 0 | 7 | 2 | 4 | 13
Platelet count decreased (Investigations) | 0 | 5 | 3 | 3 | 13
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 3 | 2 | 2 | 13
Hypotension (Vascular disorders) | 1 | 4 | 2 | 1 | 10
Sinus tachycardia (Cardiac disorders) | 0 | 3 | 2 | 2 | 7
Anorexia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 1 | 7
Fever (General disorders) | 0 | 2 | 2 | 2 | 8
Headache (Nervous system disorders) | 1 | 2 | 2 | 2 | 7
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 3 | 2 | 2 | 6
Nausea (Gastrointestinal disorders) | 1 | 4 | 0 | 2 | 7
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 5 | 3 | 2 | 1
Hypertension (Vascular disorders) | 0 | 3 | 2 | 1 | 5
Hypokalemia (Metabolism and nutrition disorders) | 0 | 3 | 1 | 4 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 5
Cytokine release syndrome (Immune system disorders) | 1 | 1 | 0 | 0 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2 | 4
Creatinine increased (Investigations) | 0 | 1 | 2 | 1 | 3
Pain (General disorders) | 0 | 1 | 2 | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 2
Edema limbs (General disorders) | 0 | 1 | 2 | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 3
Anxiety (Psychiatric disorders) | 0 | 1 | 2 | 1 | 1
Chills (General disorders) | 0 | 2 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2 | 2
Hypomagnesimia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 3
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 2 | 1 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 2 | 0 | 1 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 2 | 0 | 2
Activated partial thromboplastin time prolonged (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 3
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 2
Agitation (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 2
Alkaline phosphatase increased (Investigations) | 0 | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Abdominal distention (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
General disorders and administration site conditions - Other, Altered Handwriting (General disorders) | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
General disorders and administration site conditions - Other, Bilateral Feet Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Blurred vision (Eye disorders) | 0 | 0 | 0 | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Immune system disorders - Other, CMV Viremia Reactivation (Immune system disorders) | 0 | 0 | 0 | 0 | 1
Cognitive disorders (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Infections and infestations - Other, CoNS Bacteremia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Edema face (General disorders) | 0 | 0 | 0 | 0 | 1
Edema trunk (General disorders) | 0 | 0 | 1 | 0 | 0
Enterocolitis infection (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Esophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Infections and infestations - Other, GPR Bacteremia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Hallucinations (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
General disorders and administration site conditions - Other, Handwriting change (General disorders) | 0 | 0 | 0 | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hyperalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypothermia (General disorders) | 0 | 0 | 0 | 0 | 1
Irritability (General disorders) | 0 | 1 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Renal and urinary disorders - Other, Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, Numbness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Papulopustular rash (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other, Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal and connective tissue disorder - Other, Worsening of knee pain] (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other, Worsening of night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
General dis...General disorders and administration site conditions - Other, COVID (General disorders) | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-02): https://cdn.clinicaltrials.gov/large-docs/29/NCT03277729/Prot_SAP_000.pdf